CLINICAL TRIAL: NCT05289271
Title: A Phase 4, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, and Immunogenicity of Vaxelis™ in Healthy Children Previously Vaccinated With a 2-Dose Primary Infant Series of Either Vaxelis™ or Hexyon™
Brief Title: Safety, Tolerability, and Immunogenicity of Vaxelis™ in Children Previously Vaccinated With Vaxelis™ or Hexyon™ (V419-016)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V419-016; V419-016 (Other: Merck); 2021-004053-23 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Vaccines, Combined; Hexavalent Vaccine
MeSH Terms: interventions — Vaxelis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: V, V, V (Experimental): Participants who received a 2-dose regimen of Vaxelis™ as infants prior to enrollment will receive a Vaxelis™ booster at ~11 months of age.
  Interventions: Biological: Vaxelis™
- Group 2: H, H, V (Experimental): Participants who received a 2-dose regimen of Hexyon™ as infants prior to enrollment will receive a Vaxelis™ booster at ~11 months of age.
  Interventions: Biological: Vaxelis™

INTERVENTIONS:
Biological: Vaxelis™ — Vaxelis™ 0.5 mL sterile suspension in prefilled syringe for intramuscular administration.
  Other Names: V419

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and immunogenicity of a booster dose of Vaxelis™ (V419) given at ~11 to 13 months of age in healthy participants who were previously vaccinated with a 2-dose primary infant series of either Vaxelis™ or Hexyon™.

ELIGIBILITY:
Inclusion Criteria:

* Has received a 2-dose infant primary series of either Vaxelis™ or Hexyon™ at approximately 2 and 4 months of age

Exclusion Criteria:

* Has known or suspected impaired immunological function
* Has known or history of functional or anatomic asplenia.
* Has a known hypersensitivity to any component of the study vaccine.
* Has a known or suspected blood dyscrasia, leukemia, lymphoma of any type or other malignant neoplasm affecting the hematopoietic and lymphatic system
* Has a bleeding disorder contraindicating intramuscular vaccination
* Has a history of Hib, hepatitis B, diphtheria, tetanus, pertussis, or poliovirus infection
* Was born to a mother with a known history of hepatitis B infection
* Had a recent febrile illness (defined as rectal temperature ≥38.1°C [≥100.5°F] or axillary temperature ≥37.8°C [≥100.0°F]) occurring at or within 72 hours prior to receipt of study vaccine
* Has encephalopathy of unknown etiology, occurring within 7 days following prior vaccination with a pertussis containing vaccine
* Has an uncontrolled neurologic disorder or uncontrolled epilepsy.
* Has a health or developmental disorder that, based on the clinical judgment of the investigator, could affect evaluation of the vaccine
* Has received or is expected to receive an immunosuppressive agent
* Meets corticosteroid use criteria
* Has received any licensed, non-live vaccine within 14 days of study vaccine
* Has received any license live vaccine within 30 days of study vaccine
* Has received a blood transfusion or blood product within 6 months of study vaccine

Ages: 11 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- Germany (6):
  - Gemeinschaftspraxis Dres. Adelt, Mettlich-Lambrecht und Denneberg ( Site 0053), Bramsche, Lower Saxony
  - Kinderärztliche Gemeinschaftspraxis ( Site 0057), Wolfsburg, Lower Saxony
  - Kinder- und Jugendärzte Hürth-Park ( Site 0054), Hürth, North Rhine-Westphalia
  - Private Practice - Dr. Petri, Kinderarztpraxis ( Site 0056), Hürth, North Rhine-Westphalia
  - Gemeinschaftspraxis Matthias Donner & Dr. Martin Lüchtrath ( Site 0052), Mönchengladbach, North Rhine-Westphalia
  - Kinderärzte im Recker Park ( Site 0058), Würselen, North Rhine-Westphalia
- Italy (2):
  - A.O.U.C. Policlinico di Bari-Hygiene ( Site 0105), Bari, Apulia
  - A.O.U. Policlinico Paolo Giaccone ( Site 0102), Palermo, Sicily
- Spain (5):
  - CHUS - Hospital Clinico Universitario-Servicio de Pediatría ( Site 0001), Santiago de Compostela, La Coruna
  - Hospital Universitario La Paz-Pediatria y Enfermedades Infecciosas ( Site 0011), Madrid, Madrid, Comunidad de
  - Hospital Universitario HM Puerta del Sur-Pediatrics ( Site 0005), Madrid, Madrid, Comunidad de
  - Hospital Antequera-Pediatrics Unit ( Site 0004), Antequera, Malaga
  - Instituto Hispalense de Pediatria- IHP1 ( Site 0006), Seville, Sevilla

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Guerra A, Costantino C, Martinon-Torres F, Westerholt S, Lambeth C, Chen Z, Lumley J, Marcek T, Johnson D, Wilck M. A phase 4, open-label study to evaluate the safety and immunogenicity of DTaP5-HBV-IPV-Hib in children previously vaccinated with DTaP2-HBV-IPV-Hib or DTaP5-HBV-IPV-Hib (V419-016). Hum Vaccin Immunother. 2024 Dec 31;20(1):2310900. doi: 10.1080/21645515.2024.2310900. Epub 2024 Feb 8. PMID 38327239
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants approximately 11 to 13 months of age, (≥327 days to ≤396 days inclusive).were enrolled in this study.
Groups:
- Group 1: V, V, V: Participants who received a 2-dose regimen of Vaxelis™ as infants prior to enrollment received a Vaxelis™ booster at ~11 months of age.
- Group 2: H, H, V: Participants who received a 2-dose regimen of Hexyon™ as infants prior to enrollment received a Vaxelis™ booster at ~11 months of age.
Period: Overall Study
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Started (Allocated participants) | 86 | 82
Treated | 85 | 82
Completed | 85 | 82
Not Completed | 1 | 0
Not completed — Mistakenly allocated, untreated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: V, V, V | Group 2: H, H, V | Total
Number analyzed (Participants) | 86 | 82 | 168
Age, Continuous [Mean (Standard Deviation); unit: Days] | 348.8 (18.8) | 344.7 (16.4) | 346.8 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 77
  Male | 42 | 49 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 60 | 105
  Not Hispanic or Latino | 34 | 21 | 55
  Unknown or Not Reported | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 85 | 82 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: Solicited injection-site AEs are predefined local (at the injection/administration site) events for which the participant's legally authorized representative was specifically questioned. Participant's legally acceptable representative used a Vaccination Report Card (VRC) to report the following solicited injection-site AEs : swelling, redness (erythema), and pain/tenderness. 95% confidence intervals (CIs) were calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 5 days postvaccination
Population: All participants who received study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 85 | 82
Percentage of participants
  Injection site erythema | 52.9 [41.8 to 63.9] | 50.0 [38.7 to 61.3]
  Injection site pain | 74.1 [63.5 to 83.0] | 56.1 [44.7 to 67.0]
  Injection site swelling | 52.9 [41.8 to 63.9] | 40.2 [29.6 to 51.7]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic AE
Description: Solicited systemic AE are predefined systemic events for which the participant's legally authorized representative was specifically questioned. Participant's legally acceptable representative used a VRC to report the following solicited systemic AEs: vomiting, drowsiness (somnolence), loss of appetite, and irritability. 95% CIs were calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 5 days postvaccination
Population: All participants who received study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 85 | 82
Percentage of participants
  Decreased appetite | 43.5 [32.8 to 54.7] | 36.6 [26.2 to 48.0]
  Irritability | 77.6 [67.3 to 86.0] | 58.5 [47.1 to 69.3]
  Somnolence | 64.7 [53.6 to 74.8] | 47.6 [36.4 to 58.9]
  Vomiting | 3.5 [0.7 to 10.0] | 8.5 [3.5 to 16.8]

3. Primary Outcome: Percentage of Participants With Unsolicited AEs
Description: An unsolicited AE is an AE that was not solicited using a VRC and that is communicated by a participant's legally authorized representative who has signed the informed consent. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. 95% CIs were calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 15 days postvaccination
Population: All participants who received study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 85 | 82
Percentage of participants | 97.6 [91.8 to 99.7] | 92.7 [84.8 to 97.3]

4. Primary Outcome: Percentage of Participants With a Serious AE (SAE)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. 95% CIs were calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 40 days postvaccination
Population: All participants who received study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 85 | 82
Percentage of participants | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.6]

5. Primary Outcome: Percentage of Participants With Diphtheria Toxoid Antibodies ≥0.1 IU/mL
Description: Human antibodies to diphtheria toxoid were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with the lower limit of quantitation (LLOQ) for diphtheria antibody of 0.005 IU/mL. The percentage of participants with diphtheria toxoid antibodies ≥0.1 international units per milliliter (IU/mL) one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: All enrolled participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint. Potential deviations include, but are not limited to failure to receive study vaccine at Visit 1 (Day 1); receipt of a prohibited medication or prohibited vaccine within the study window; or collection of blood sample at Visit 2 outside the prespecified window (Day 26 to Day 40).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 69 | 74
Percentage of participants | 100.0 [94.8 to 100.0] | 98.6 [92.7 to 100.0]

6. Primary Outcome: Percentage of Participants With Tetanus Toxoid Antibodies ≥0.1 IU/mL
Description: Human antibodies to tetanus toxoid were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with a LLOQ for tetanus antibody of 0.01 IU/mL. The percentage of participants with tetanus toxoid antibodies ≥0.1 IU/mL one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 69 | 74
Percentage of participants | 98.6 [92.2 to 100.0] | 98.6 [92.7 to 100.0]

7. Primary Outcome: Percentage of Participants With Pertussis Toxoid (PT) Vaccine Response
Description: Human antibodies to pertussis toxoid were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with a LLOQ for pertussis antibody of 2.00 EU/mL. The percentage of participants meeting response criteria for PT is based on pre-vaccination level of PT is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 64 | 71
Percentage of participants | 98.4 [91.6 to 100.0] | 94.4 [86.2 to 98.4]

8. Primary Outcome: Percentage of Participants With Filamentous Hemagglutinin (FHA) Vaccine Response
Description: Human antibodies to FHA were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with a LLOQ for FHA antibody of 2.00 EU/mL. The percentage of participants meeting response criteria for FHA response will be based on pre-vaccination level of FHA. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 64 | 71
Percentage of participants | 98.4 [91.6 to 100.0] | 90.1 [80.7 to 95.9]

9. Primary Outcome: Percentage of Participants With Haemophilus Influenzae Type b Polyribosylribitol Phosphate (Hib-PRP) Antibodies ≥1.0 µg/mL
Description: Human antibodies to Hib-PRP were quantified using the Vacczyme™ Human Anti-Haemophilus influenzae Type b Enzyme Immunoassay Kit. Levels of anti-Hib IgG were quantified by interpolation from a standard curve that has been calibrated to the FDA lot 1983 reference serum. The percentage of participants with Hib-PRP antibodies ≥0.1 IU/mL one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 73 | 76
Percentage of participants | 89.0 [79.5 to 95.1] | 90.8 [81.9 to 96.2]

10. Primary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Antibodies ≥10 mIU/mL
Description: Human antibodies to HBsAg were quantified using an Enhanced Chemiluminescence (ECi) assay, with the hepatitis B WHO International reference standard at 10 mIU/mL as a control in every assay, and the LLOQ of the assay is 5 mIU/mL. The percentage of participants with HBsAg antibodies ≥10 milli-international per liter (mIU/mL) one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 56 | 69
Percentage of participants | 100.0 [93.6 to 100.0] | 94.2 [85.8 to 98.4]

11. Primary Outcome: Percentage of Participants With Poliovirus Serotype 1 Neutralizing Antibodies (Nab) ≥1:8 Dilution
Description: Human antibodies to poliovirus serotype 1 were quantified with a neutralization assay by utilizing Vero cells and wild type poliovirus strain 1 as the challenge virus. The Karber method was used to determine the serum dilution that neutralized 50% of the challenge virus, with results expressed as titers (1:dilution), and the LLOQ was 1:4. dilution. The percentage of participants with poliovirus serotype 1 Nab ≥1:8 dilution one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 66 | 69
Percentage of participants | 100.0 [94.6 to 100.0] | 95.7 [87.8 to 99.1]

12. Primary Outcome: Percentage of Participants With Poliovirus Serotype 2 Neutralizing Antibodies (Nab) ≥1:8 Dilution
Description: Human antibodies to poliovirus serotype 2 were quantified with a neutralization assay by utilizing Vero cells and wild type poliovirus strain 2 as the challenge virus. The Karber method was used to determine the serum dilution that neutralized 50% of the challenge virus, with results expressed as titers (1:dilution), and the LLOQ was 1:4. dilution. The percentage of participants with poliovirus serotype 2 Nab ≥1:8 dilution one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 66 | 69
Percentage of participants | 100.0 [94.6 to 100.0] | 100.0 [94.8 to 100.0]

13. Primary Outcome: Percentage of Participants With Poliovirus Serotype 3 Neutralizing Antibodies (Nab) ≥1:8 Dilution
Description: Human antibodies to poliovirus serotype 3 were quantified with a neutralization assay by utilizing Vero cells and wild type poliovirus strain 3 as the challenge virus. The Karber method was used to determine the serum dilution that neutralized 50% of the challenge virus, with results expressed as titers (1:dilution), and the LLOQ was 1:4. dilution. The percentage of participants with poliovirus serotype 3 Nab ≥1:8 dilution one month after Vaxelis™ as the 3rd dose of a vaccination series is presented. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 66 | 69
Percentage of participants | 97.0 [89.5 to 99.6] | 100.0 [94.8 to 100.0]

14. Secondary Outcome: Percentage of Participants With Pertactin (PRN) Vaccine Response
Description: Human antibodies to PRN were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with a LLOQ for PRN of 2.00 EU/mL.The percentage of participants meeting response criteria for PRN was based on pre-vaccination level of PRN. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 64 | 71
Percentage of participants | 92.2 [82.7 to 97.4] | 22.5 [13.5 to 34.0]

15. Secondary Outcome: Percentage of Participants With Fimbriae 2/3 (FIM 2/3) Vaccine Response
Description: Human antibodies to FIM 2/3 were quantified using the Meso Scale Discovery Electrochemiluminescence serological assay based on an established reference standard sample curve with a LLOQ for pertussis antibody of 2.00 EU/mL.
  The percentage of participants meeting response criteria for FIM 2/3 was based on pre-vaccination level of FIM 2/3. The 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: 30 days postvaccination (at ~12 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
Number analyzed (Participants) | 64 | 71
Percentage of participants | 95.3 [86.9 to 99.0] | 69.0 [56.9 to 79.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs): from vaccination up to 40 days post-vaccination; All-cause mortality (ACM): From allocation up to 40 days post-vaccination
Description: AE population: All participants who received study vaccination. ACM population: all allocated participants.
Arm/Group | Group 1: V, V, V | Group 2: H, H, V
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/85 | 1/82
Other Adverse Events (participants affected / at risk) | 83/85 | 75/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: V, V, V (N=85) | Group 2: H, H, V (N=82)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: V, V, V (N=85) | Group 2: H, H, V (N=82)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5) | 8 (8)
Injection site erythema (General disorders) | 45 (45) | 41 (41)
Injection site induration (General disorders) | 0 (0) | 6 (6)
Injection site pain (General disorders) | 63 (63) | 46 (46)
Injection site swelling (General disorders) | 45 (45) | 33 (33)
Pyrexia (General disorders) | 34 (35) | 40 (47)
Decreased appetite (Metabolism and nutrition disorders) | 37 (38) | 30 (31)
Somnolence (Nervous system disorders) | 55 (55) | 39 (42)
Irritability (Psychiatric disorders) | 66 (66) | 48 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT05289271/Prot_SAP_000.pdf